CLINICAL TRIAL: NCT04641819
Title: Yangzheng Compound Mixture in the Treatment of Sleep Disorder in Cancer Patients With Qi-Yin Deficiency Syndrome During Chemotherapy: a Multicenter, Randomized, Prospective, Real-world Study
Brief Title: Yangzheng Compound Mixture in the Treatment of Sleep Disorder in Cancer Patients
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: ShuGuang Hospital (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry); Shaanxi Buchang Pharmaceutical Co., Ltd (Industry)
Responsible Party: Principal Investigator, Qi Li, Professor, ShuGuang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESPRESSO
Record Dates: First submitted 2020-11-06; First posted 2020-11-24 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Carcinoma; Sleep Disorder
Keywords: Yangzheng Compound Mixture; Carcinoma; Sleep Disorder
MeSH Terms: conditions — Carcinoma; Sleep Wake Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yangzheng Compound Mixture plus conventional treatment (Experimental): Yangzheng Compound Mixture: 10mL, 2 doses each time, 3 times a day, three weeks for a course of treatment. Investigators recommended that the participants of experimental group should use Yangzheng Compound Mixture for 2 courses at least.
  Conventional treatment:
  Antitumor therapies: chemotherapy or combined chemotherapy. Sleep disorders: includes but is not limited to pharmacotherapy and exercise therapy.
  The examination, diagnosis and treatment of other concomitant diseases and tumor complications are based on clinical routine. We will collect information about all the combined medicine.
  Interventions: Drug: Yangzheng Compound Mixture; Other: Conventional Treatment
- conventional treatment only (Other): Antitumor therapies: chemotherapy or combined chemotherapy. Sleep disorders: includes but is not limited to pharmacotherapy and exercise therapy.
  The examination, diagnosis and treatment of other concomitant diseases and tumor complications are based on clinical routine. We will collect information about all the combined medicine.
  Interventions: Other: Conventional Treatment

INTERVENTIONS:
Drug: Yangzheng Compound Mixture — At the end of the treatment period, the investigator can decide whether to continue the medication based on the improvement of the subjects' sleep disturbance.
  Medication during the follow-up period: subjects will enter the follow-up period after completing one course of Yangzheng Compound Mixture treatment or the end of the treatment period. Visits will be conducted once every 3 weeks, at least 2 times and no more than 4 times. For subjects in the experimental group, doctors can decide whether the patients should continue to receive Yangzheng Compound Mixture therapy in the follow-up period according to the improvement of sleep disorders, while for subjects in the control group, the patients can choose to start receiving Yangzheng Compound Mixture therapy in the follow-up period according to their own wishes and doctors' suggestions.
  Other Names: Z10970042（NMPA Approval Number）
  Arms: Yangzheng Compound Mixture plus conventional treatment
Other: Conventional Treatment — Including treatment of sleep disorders and tumor which shall follow the clinical guidelines.

SUMMARY:
This is a nationwide, multicenter, randomized, prospective, real-world study. The purpose of this study is to evaluate the effect and safety of Yangzheng Compound Mixture in the treatment of sleep disorder in cancer patients with Qi-Yin deficiency syndrome during chemotherapy.

DETAILED DESCRIPTION:
Sleep disturbance is one of the most common symptoms in cancer patients, the morbidity is about 60%. Drugs commonly used to treat sleep disorders include benzodiazepines, hypnotic antidepressants and melatonin receptors agonists. The short-term efficacy of these drugs has been proven in many clinical trials, but long-term medications bear the risk of adverse reactions and addiction.

Yangzheng Compound Mixture is an extract of several traditional Chinese medicines, used as a basic prescription for cancer therapy, especially for patients who received chemotherapy with Qi-Yin deficiency syndrome, which often lead to sleep disturbance, fatigue and anorexia. According to some clinical and basic studies, Yangzheng Compound Mixture also has antitumor and immunomodulatory effects.

In this study, about 10 research centers will participate. We planned to enroll 1526 cancer patients (1144 cases in the observation group and 382 cases in the control group) with Qi-Yin deficiency Syndrome and sleep disorders during the period of receiving chemotherapy or combination of chemotherapy. The dynamic random method was adopted in this study, participants will be randomly divided into the experimental group (Yangzheng Compound Mixture plus conventional treatment) and control group (conventional treatment only), all of them will be interviewed once every 3 weeks until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18;
* Histologically or cytologically confirmed as malignant tumor;
* Receiving chemotherapy or a combination of chemotherapy;
* The syndrome differentiation of traditional Chinese medicine is the Qi-yin deficiency syndrome;
* Sleep disorders were diagnosed by investigators and the Pittsburgh Sleep Quality Index (PSQI) score was ≥ 8;
* The date of diagnosis of sleep disorder is later than the date of the first diagnosis of cancer. Or patients with sleep disorders for a long time receiving regular treatment，sleep disorders aggravated after cancer diagnosis or chemotherapy;
* Pain has been controlled well [patients were being treated with analgesics regularly，numerical rating scale（NRS） score ≤ 3];
* The participant must be able to read and express themselves clearly, can communicate with investigators and cooperate in completing the questionnaire;
* Participants voluntarily join the study with good compliance, and are willing to sign a written informed consent document;
* Survival period will be longer than 6 months.

Exclusion Criteria:

* Pregnant or lactating women;
* Allergic to Yangzheng Compound Mixture;
* Previous diagnosis of sleep apnea;
* The laboratory test value of liver and renal function is more than 2.5 times the upper limit of normal value;
* Symptoms of brain metastasis due to malignant tumor has not been effectively controlled;
* Participating in other drug clinical trials which did not allow to participate in this study;
* Refused to cooperate with follow-up;
* The researchers did not consider it appropriate for the patients to participate in this study for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1127 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Best effective rate for sleep disorder treatment | Measurement was taken at week 6.
  Proportion of participants with a minimum PSQI score < 8 during the treatment period.
Effective rate for sleep disorder treatment | Measurement was taken at week 6.
  Proportion of participants with PSQI score < 8 after the end of the different treatment courses.
Improvement rate for sleep disorder treatment | Measurement was taken at week 6.
  Proportion of participates whose PSQI score decreased during treatment compared with the baseline.
Change of PSQI score compared with baseline | Baseline and week 6.
  The PSQI score difference between the end of different treatment courses and baseline.
Score of Pittsburgh Sleep Quality Index (PSQI), Sleep duration, Sleep efficiency, Subjective sleep quality, Sleep latency. | Measurement was taken at week 6.
  1. The outcomes were evaluated using the PSQI scale.
  2. Sleep duration: response to question 4;
  3. Sleep efficiency= (hours slept/ hours in bed) * 100%; Hours slept: response to question 4; Hours in bed: calculated from responses to questions 1 and 3;
  4. Subjective sleep quality: response to question 9;
  5. Sleep latency: response to question 2.
Incidence and severity of AE or SAE | Start of treatment until 30 days after the last day of the sleep disorder treatment
  AE: Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
  SAE: A serious adverse event (experience) or reaction is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
Incidence and severity of ADR or SADR | Start of treatment until 30 days after the last day of the sleep disorder treatment
  All noxious and unintended responses to a medicinal product related to any dose should be considered adverse drug reactions. A SADR is a serious ADR according to the above criteria of SAE.

SECONDARY OUTCOMES:
Use frequency of hypnotic agents | Up to 18 weeks since the start of treatment
  Response to question 6 of the PSQI scale.
Appetite | Up to 18 weeks since the start of treatment
  Appetite was evaluated by using the Cancer Appetite and Symptom Questionnaire(CASQ).
Fatigue | Up to 18 weeks since the start of treatment
  Fatigue was evaluated by using the Brief Fatigue Inventory(BFI).
Quality of life (QOL) | Up to 18 weeks since the start of treatment
  Quality of Life (QOL) was measured by using the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30).
Traditional Chinese Medical symptoms scale | Up to 18 weeks since the start of treatment
  Traditional Chinese Medical (TCM) symptoms were measured from these six aspects: weakness, shortness of breath, palpitations, deficiency-heat and vexation, dry mouth, sweat. The minimum score is 0 and the maximum value is 18. Higher scores of TCM scale means a worse outcome.

OTHER OUTCOMES:
Proportion of leukocyte-increasing drugs used | Up to 18 weeks since the start of treatment
  Proportion of participates used leukocyte-increasing medication during the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Qi Li, PhD, Principal Investigator — Shuguang Hospital Affiliated with Shanghai University of TCM
Locations (10):
- China (10):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - First Affiliated Hospital, Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang
  - Jiamusi Cancer Hospital, Jiamusi, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The Second Affiliated Hospital of Hunan University of Chinese Medicine, Changsha, Hunan
  - The Third Affiliated Hospital of Shandong First Medical University, Jinan, Shandong
  - Shuguang Hospital Affiliated with Shanghai University of TCM, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Affiliated Hospital of Shanxi University of Chinese Medicine, Xianyang, Shanxi
  - Cancer Hospital of The University of Chinese Academy of Sciences, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No